CLINICAL TRIAL: NCT02556554
Title: A Single-center, Prospective, 'Open-label,' Investigator-initiated Pilot Study Evaluating the Role of Continuous Glucose Monitor (CGM) Use Either Alone or With Remote Monitoring Capabilities in Pregnancy Associated With Type 1 Diabetes
Brief Title: Pilot Prospective CGM Quality Improvement (QI) Project in Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: DexCom, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-1006
Record Dates: First submitted 2015-09-11; First posted 2015-09-22 (Estimated); Results first posted 2020-07-21 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Diabetes Mellitus, Type I
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Routine Care (No Intervention): Standard of Care in the Pregnancy and Women's Health clinic.
- Dexcom G4 Platinum CGM system (Active Comparator): An intervention arm using the Dexcom G4 or G5 Platinum® CGM system during pregnancy.
  Interventions: Device: Dexcom G4 or G5 Platinum CGM system
- Dexcom G4 Platinum CGM system with Share™ (Active Comparator): A treatment arm using the Dexcom G4 or G5 Platinum® CGM system with Share™ remote monitoring capabilities during pregnancy.
  Interventions: Device: Dexcom G4 or G5 Platinum CGM system with Share

INTERVENTIONS:
Device: Dexcom G4 or G5 Platinum CGM system — Intervention arm using the Dexcom G4 or G5 Platinum® CGM system during pregnancy
  Arms: Dexcom G4 Platinum CGM system
Device: Dexcom G4 or G5 Platinum CGM system with Share — Treatment arm using the Dexcom G4 or G5 Platinum® CGM system with Share™
  Arms: Dexcom G4 Platinum CGM system with Share™

SUMMARY:
A single-center, prospective, 'open-label,' investigator-initiated pilot study evaluating the role of continuous glucose monitor (CGM) use either alone or with remote monitoring capabilities during pregnancy associated with T1DM.

DETAILED DESCRIPTION:
A single-center, prospective, 'open-label,' investigator-initiated pilot study evaluating the role of continuous glucose monitor (CGM) use either alone or with remote monitoring capabilities that enable subjects to share CGM data with family and friends (whom the investigators will call "followers" in this protocol) among women with T1DM associated with pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent before any study-related activities
* Female aged 18 years and older
* T1D duration >1 year
* Pregnancy with confirmation of gestational age 13 weeks or less
* Willingness to routinely practice at least 3-7 blood glucose measurements per day
* Using MDI or CSII therapy
* Willingness to provide an A1C level
* Ability and willingness to adhere to the protocol including scheduled study visits for the duration of the pregnancy
* Able to speak, read, and write English

Exclusion Criteria

* Extensive skin changes/diseases that inhibit wearing a sensor on normal skin
* Known allergy to adhesives
* Any other condition, as determined by the investigator, which could make the subject unsuitable for the trial, impairs the subject's suitability for the trial, or impairs the validity of the informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2015-08; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarit Polsky, MD, MPH, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Aurora, Colorado, United States

REFERENCES:
- [Derived] Shah VN, Snell-Bergeon JK, Demmitt JK, Joshee P, Garcetti R, Pyle L, Polsky S. Relationship Between Time-in-Range, HbA1c, and the Glucose Management Indicator in Pregnancies Complicated by Type 1 Diabetes. Diabetes Technol Ther. 2021 Dec;23(12):783-790. doi: 10.1089/dia.2021.0093. Epub 2021 Nov 3. PMID 34524020
- [Derived] Buschur EO, Campbell K, Pyle L, Garcetti R, Joshee P, Demmitt JK, Snell-Bergeon JK, Polsky S. Exploratory Analysis of Glycemic Control and Variability Over Gestation Among Pregnant Women with Type 1 Diabetes. Diabetes Technol Ther. 2021 Nov;23(11):768-772. doi: 10.1089/dia.2021.0138. PMID 34115946
- [Derived] Polsky S, Garcetti R, Pyle L, Joshee P, Demmitt JK, Snell-Bergeon JK. Continuous Glucose Monitor Use With Remote Monitoring Reduces Fear of Hypoglycemia in Pregnant Women With Type 1 Diabetes: A Pilot Study. J Diabetes Sci Technol. 2020 Jan;14(1):191-192. doi: 10.1177/1932296819890864. Epub 2019 Nov 28. No abstract available. PMID 31779476

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From 08/2015 to 06/2016, investigators enrolled women in preconception and the 1st trimester at the Barbara Davis Center, and followers. Other women consented for the retrospective (no CGM) group. Follower data only included answers to monthly questionnaires. Study registration was delayed due to staffing issues and account set-up in the system.
Pre-assignment Details: Study cohorts: (1) women with T1D prospectively enrolled in 1st trimester or when planning pregnancy, (2) followers (family/friends) of women in the 1st cohort, and (3) women with T1D with a pregnancy within the past 3 years who did not use CGM therapy during gestation (retrospective). Follower data only included answers to monthly questionnaires.
Groups:
- Followers for Dexcom Alone: Followers of Pregnant Women Using Dexcom Alone
- Followers for Dexcom Share: Followers of Pregnant Women Using Dexcom with Share
Period: Overall Study
Arm/Group | Routine Care | Dexcom G4 Platinum CGM System | Dexcom G4 Platinum CGM System With Share™ | Followers for Dexcom Alone | Followers for Dexcom Share
Started | 8 | 14 | 19 | 12 | 14
Completed | 8 | 13 | 15 | 12 | 14
Not Completed | 0 | 1 | 4 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline demographics data was not collected for the two "Followers" arms consisting of family/friends of the persons in the "Dexcom G4 Platinum CGM System" and "Dexcom G4 Platinum CGM System With Share™" arms.
Groups:
- Total: Total of all reporting groups
Arm/Group | Routine Care | Dexcom G4 Platinum CGM System | Dexcom G4 Platinum CGM System With Share™ | Total
Number analyzed (Participants) | 8 | 13 | 15 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 13 | 15 | 36
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 27.6 [20.7 to 29.5] | 24.4 [21.2 to 30.3] | 28.9 [26.7 to 31.0] | 27.3 [23.5 to 30.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 13 | 15 | 36
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Race/ethnicity data were not obtained from retrospective chart review (no CGM) group.
  Participants
    Race/ethnicity: number analyzed (Participants) | 0 | 13 | 15 | 28
    Race/ethnicity: Caucasian |  | 8 | 14 | 22
    Race/ethnicity: Hispanic/Latina |  | 3 | 1 | 4
    Race/ethnicity: Asian/Oriental |  | 1 | 0 | 1
    Race/ethnicity: Other |  | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 8 | 13 | 15 | 36
Method of insulin delivery, n (%) [Count of Participants; unit: Participants]
  Multiple daily injections (MDI) | 4 | 7 | 2 | 13
  Continuous subcutaneous insulin infusion (CSII) | 3 | 6 | 13 | 22
  Unknown | 1 | 0 | 0 | 1
Preconception hemoglobin A1C (%) [Median (Inter-Quartile Range); unit: %] | 7.2 [5.5 to 8.4] | 8.1 [7.2 to 9.0] | 7.1 [6.3 to 8.4] | 7.4 [6.6 to 8.7]

OUTCOME MEASURES:

1. Primary Outcome: Changes in Glucose Variability
Description: Glucose variability as measured by glucose excursions from CGM
Time Frame: From first pregnancy visit to delivery
Population: CGM metrics among CGM Share and CGM Alone (not among no CGM since they did not use a CGM)
Measure: Median (Inter-Quartile Range); unit: % time spent in range
Arm/Group | Dexcom G4 Platinum CGM System | Dexcom G4 Platinum CGM System With Share™
Number analyzed (Participants) | 13 | 15
% time spent in range
  Time spent <65 mg/dL (1st trimester) | 7.5 [4.7 to 9.0] | 7.3 [3.6 to 8.2]
  Time spent 65-140 mg/dL (1st trimester) | 52.8 [46.4 to 73.0] | 59.8 [54.5 to 68.7]
  Time spent >140 mg/dL (1st trimester) | 38.2 [21.7 to 49.0] | 35.1 [24.3 to 41.0]
  Time spent <65 mg/dL (2nd trimester) | 5.0 [3.8 to 7.5] | 5.3 [4.0 to 8.4]
  Time spent 65-140 mg/dL (2nd trimester) | 50.7 [43.6 to 61.8] | 56.6 [48.7 to 69.0]
  Time spent >140 mg/dL (2nd trimester) | 44.2 [27.8 to 51.7] | 37.2 [21.9 to 43.1]
  Time spent <65 mg/dL (3rd trimester) | 4.0 [3.6 to 4.6] | 4.5 [3.4 to 6.1]
  Time spent 65-140 mg/dL (3rd trimester) | 53.5 [42.6 to 59.4] | 62.3 [49.9 to 70.4]
  Time spent >140 mg/dL (3rd trimester) | 43.2 [35.4 to 52.8] | 34.4 [23.1 to 46.8]

2. Primary Outcome: Change(s) in Behavior and/or Concerns of Diabetics.
Description: Change(s) in behavior and/or concerns of diabetics as detected by the hypoglycemia fear questionnaire. Behavior sub-scale score ranges from 10-50, with higher scores indicating more behavioral changes in the participant's daily routine to avoid low blood sugar. Worry sub-scale score ranges from 17-85, with higher scores indicating more worry or concerns because of low blood sugar. Total score ranges from 27-135, with higher scores for both sub-scales indicating more fear and a worse outcome.
Time Frame: From first pregnancy visit to delivery
Population: Hypoglycemia Fear Survey results (higher scores indicate more behavioral changes, worry, or total fear scores). Only prospectively enrolled pregnant women were administered this questionnaire (CGM Alone and CGM Share groups).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dexcom G4 Platinum CGM System | Dexcom G4 Platinum CGM System With Share™
Number analyzed (Participants) | 13 | 15
score on a scale
  Behavior score (1st trimester) | 28.8 (5.8) | 27.9 (3.9)
  Worry Score (1st Trimester) | 45.1 (14.8) | 34.0 (7.2)
  Total Score (1st Trimester) | 73.8 (14.1) | 61.9 (9.4)
  Behavior score (2nd trimester) | 28.2 (6.9) | 28.9 (4.5)
  Worry Score (2nd Trimester) | 37.5 (12.5) | 34.6 (9.7)
  Total Score (2nd Trimester) | 65.8 (15.4) | 63.4 (13.0)
  Behavior score (3rd trimester) | 28.6 (6.6) | 28.2 (4.1)
  Worry Score (3rd Trimester) | 43.4 (19) | 37.4 (7.8)
  Total Score (3rd Trimester) | 72.0 (23.8) | 65.5 (10.7)

3. Secondary Outcome: Change in A1C.
Description: Change in A1C with CGM alone and CGM with Share™ compared to no CGM use.
Time Frame: From first pregnancy visit to delivery
Population: Least squares mean HbA1c by group in a model without interaction and without adjustment for preconception HbA1c.
Measure: Least Squares Mean (Standard Error); unit: HbA1C %
Arm/Group | Routine Care | Dexcom G4 Platinum CGM System | Dexcom G4 Platinum CGM System With Share™
Number analyzed (Participants) | 8 | 13 | 15
HbA1C % | 6.85 (0.13) | 6.84 (0.09) | 6.19 (0.07)

4. Secondary Outcome: Evaluation of Maternal and Fetal Outcomes.
Description: Evaluation of Maternal and fetal outcomes (eclampsia/pre-eclampsia, live birth rates, birth weight, neonatal hypoglycemia, and other similar measures)
Time Frame: From first pregnancy visit to delivery
Population: Maternal and fetal outcomes among prospective pregnant study arms (CGM Share and CGM Alone)
Measure: Count of Participants; unit: Participants
Arm/Group | Dexcom G4 Platinum CGM System | Dexcom G4 Platinum CGM System With Share™
Number analyzed (Participants) | 13 | 15
Participants
  Cesarean section, n (%) | 8 | 13
  Preeclampsia, n (%) | 4 | 4
  <37 weeks gestation at delivery, n (%) | 7 | 4
  Large-for-gestational age infant, n (%) | 5 | 8
  Macrosomia, n (%) | 0 | 3
  Small-for-gestational age infant, n (%) | 0 | 1
  Neonatal hypoglycemia, n (%) | 7 | 11
  Neonatal jaundice, n (%) | 8 | 5
  Neonatal hypoxemia, n (%) | 6 | 1
  Neonatal intensive care unit admission, n (%) | 5 | 7
  Progression of diabetic retinopathy (both eyes) | 2 | 2
  Progression of diabetic retionpathy (one eye) | 3 | 2
  Progression of diabetic retinopathy (neither eye) | 5 | 4

ADVERSE EVENTS:
Time Frame: Pregnancy and up the the first 6 weeks post-partum, an average of 1 year, for prospectively enrolled study arms (CGM Share and CGM Alone)
Description: Severe hypoglycemia was defined as glucose <70 mg/dL requiring the assistance of a third party. Miscarriage was defined as 1st trimester fetal loss (women who miscarried and became pregnant again during the enrollment period could re-enroll). Number at risk for miscarriage includes all pregnancies, but number at risk for mortality includes participants (not individual pregnancies). Adverse events were captured and recorded only in prospectively enrolled arms (does not include no CGM group).
Groups:
- Followers of Dexcom G4 Platinum CGM System: Followers (family or friends) of Dexcom G4 Platinum CGM system
- Followers of Dexcom G4 Platinum CGM System With Share™: Followers (family or friends) of Dexcom G4 Platinum CGM system with Share™
Arm/Group | Dexcom G4 Platinum CGM System | Dexcom G4 Platinum CGM System With Share™ | Followers of Dexcom G4 Platinum CGM System | Followers of Dexcom G4 Platinum CGM System With Share™
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/15 | 0/12 | 0/14
Serious Adverse Events (participants affected / at risk) | 3/13 | 4/15 | 0/12 | 0/14
Other Adverse Events (participants affected / at risk) | 0/13 | 0/15 | 0/12 | 0/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dexcom G4 Platinum CGM System (N=13) | Dexcom G4 Platinum CGM System With Share™ (N=15) | Followers of Dexcom G4 Platinum CGM System (N=12) | Followers of Dexcom G4 Platinum CGM System With Share™ (N=14)
severe hypoglycemic episode (Endocrine disorders) | 0 (0) | 2 (3) | NA | NA — Severe hypoglycemia was defined as hypoglycemia (glucose <70 mg/dL) requiring the assistance of a third party.
Miscarriage (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 2 (2) | NA | NA — Fetal loss within the 1st trimester

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-17): https://cdn.clinicaltrials.gov/large-docs/54/NCT02556554/Prot_SAP_000.pdf